CLINICAL TRIAL: NCT04427618
Title: Tranexamic Acid in the Prevention of Postpartum Hemorrhage in Elective Caesarean Section: a Randomised Controlled Trial
Brief Title: Tranexamic Acid in the Prevention of Postpartum Hemorrhage in Elective Caesarean Section
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2019/2425
Record Dates: First submitted 2020-06-07; First posted 2020-06-11 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2021-08

CONDITIONS: Postpartum Hemorrhage; Tranexamic Acid
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Intravenous 1g TXA (500mg/5ml, given intermittent over approximately 10 minutes) given within approximately 10 minutes before skin incision, and Intravenous oxytocin 5 units post delivery of the baby.
  Interventions: Drug: Tranexamic acid
- Control group (Placebo Comparator): Intravenous 10ml normal saline (placebo) given within approximately 10 minutes before skin incision, and intravenous oxytocin 5 units post delivery of the baby
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Tranexamic acid — Intravenous 1g TXA (500mg/5ml, given intermittent over approximately 10 minutes) given within approximately 10 minutes before skin incision
  Arms: Intervention group
Drug: Normal saline — Intravenous 10ml normal saline (placebo) given within approximately 10 minutes before skin incision
  Arms: Control group

SUMMARY:
In obstetrics, postpartum haemorrhage (PPH) continues to be a major contributor to maternal morbidity and mortality worldwide. Uterine atony is the most common cause of PPH, and the prophylactic use of uterotonics, specifically oxytocin, is the standard of care for PPH prophylaxis. It is believed that tranexamic acid (TXA) can enhance the hemostatic process further by inhibiting the fibrinolytic system.

TXA is an antifibrinolytic that has been studied in many different patient population for its use in reducing blood loss ranging from gynaecological and non gynaecological surgeries, to trauma patients. It has been found to reduce mortality in treatment of patients with PPH, and recent evidence have found promising results in its use for prophylaxis of PPH.

ELIGIBILITY:
Inclusion Criteria:

* All English speaking patients
* Above 21 year old
* Undergoing elective caesarean section.

Exclusion Criteria:

* Known/suspected placenta accreta antenatally
* Contraindications to syntocinon and tranexamic acid such as hypersensitivity to these medications
* Known thrombophilia or coagulopathy
* History of thromboembolic events
* Severe cardiac/renal/liver disease
* Poorly controlled hypertension /severe preeclampsia (BP > 160/100)/eclampsia

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2021-10-03 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Estimated blood loss | Intraoperative
  This will be calculated estimated blood loss, defined as estimated blood volume x (preoperative hematocrit - postoperative hematocrit) ÷ preoperative hematocrit. Estimated blood volume in milliliters was calculated by body weight in kilograms x 85.

SECONDARY OUTCOMES:
Change in hemoglobin and hematocrit level | Preoperative to 48 hours postoperative
  Comparison of full blood count results prior to surgery and within approximately 48 hours post surgery
Need for additional medical intervention including blood transfusion, additional uterotonics | During surgery and up to 3 days after surgery
Incidence of postpartum hemorrhage: defined as >1000ml total blood loss within 24 hours after delivery | During surgery and up to 24 hours from surgery
Maternal thrombotic event such as deep vein thrombosis and pulmonary embolism | Intraoperative to 4 weeks post surgery
  Patients will be reviewed for signs and symptoms of thromboembolic events. They will be reviewed daily post surgery in the ward as per routine protocol. Generally, all post caesarean section patients will be warded till post operative day 3. They will also have a routine follow up 4 weeks post surgery.
Neonatal APGAR score | At delivery
  Neonatal APGAR score at 1 and 5 minutes of life
Neonatal birth weight | At delivery
Neonatal admission to special care nursery or intensive care unit | At delivery
Diagnosis of thromboembolic events in the neonate | Up to 4 weeks post delivery
Gravimetric estimation of blood loss during the surgery | Intraoperative
  This would be assessed by weighing the swabs and drapes as well as measuring the volume of suction aspirated once the amniotic fluid volume had been deducted
Provider estimated blood loss | Intraoperative
  Estimated by the surgical team

CONTACTS AND LOCATIONS:
Overall Officials: Manisha Mathur, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided